CLINICAL TRIAL: NCT06117605
Title: Protocol for a Pragmatic, Multicenter, Factorial, Randomized Controlled Trial of Sepsis Electronic Prompting for Timely Intervention and Care (SEPTIC Trial) for Emergency Department Patients
Brief Title: Sepsis Electronic Prompting for Timely Intervention and Care for Emergency Department Patients
Acronym: SEPTIC-ED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Jason Adelman, Associate Professor of Medicine, Columbia University
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Health Services Research
Other Study IDs: AAAU1002 - ED
Record Dates: First submitted 2023-10-31; First posted 2023-11-07 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-08

CONDITIONS: Sepsis; Electronic Health Records; Clinical Decision Support Systems
Keywords: sepsis; alerts; clinical decision support systems; informatics; health information technology
MeSH Terms: conditions — Sepsis

STUDY DESIGN:
Intervention Model Description: If a patient is randomized to a group without an alert, the alert will instead be a hidden "silent" alert that does not display. However, a timestamp of when the alert was triggered is still recorded even though the alert did not display. This timestamp is used for the primary and secondary outcomes.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Care providers will be unblinded in that nurses and clinicians will be aware if they receive an alert for the patient.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- No alert (No Intervention): Participants will receive no physician alert or registered nurse (RN) alert.
- Nurse alert (Experimental): Participants will receive RN alert.
  Interventions: Other: Nurse SIRS alert
- Prescribing clinician alert (Experimental): Participants will receive physician alert.
  Interventions: Other: Prescribing clinician SIRS alert
- Nurse alert and prescribing clinician alert (Experimental): Participants will receive physician alert and RN alert.
  Interventions: Other: Nurse SIRS alert; Other: Prescribing clinician SIRS alert

INTERVENTIONS:
Other: Nurse SIRS alert — An electronic alert will display when a nurse opens the patient chart of a patient who meets SIRS criteria.
  Arms: Nurse alert; Nurse alert and prescribing clinician alert
Other: Prescribing clinician SIRS alert — An electronic alert will display when a prescribing clinician opens the patient chart of a patient who meets SIRS criteria.
  Arms: Nurse alert and prescribing clinician alert; Prescribing clinician alert

SUMMARY:
The goal of this clinical trial is to study systemic inflammatory response syndrome (SIRS) electronic health record (EHR) alerts for sepsis in the emergency department (ED). The main question it aims to answer is: do nurse alerts, prescribing clinician alerts, or both nurse and prescribing clinician alerts improve time to sepsis treatment for patients in the ED?

Nurses and prescribing clinicians will receive SIRS alerts based on the group to which the patient is randomly assigned. Researchers will compare four groups: no alerts, nurse alerts only, prescribing clinician alerts only, or both nurse and prescribing clinician alerts.

DETAILED DESCRIPTION:
SEPTIC is a master protocol for two trials on distinct subpopulations: emergency department (ED) patients and inpatients. This protocol "ID: AAAU1002 - ED" describes the ED subpopulation study while "ID: AAAU1002 - IP" describes the inpatient subpopulation study.

Sepsis is a major cause of death both globally and in the United States. Early identification and treatment of sepsis are crucial for improving outcomes. International guidelines recommend hospital sepsis screening programs, which are commonly implemented in the electronic health record (EHR) as an interruptive screening alert based on systemic inflammatory response syndrome (SIRS) criteria. Despite widespread use, it is unknown whether these sepsis screening and alert tools improve the delivery of high-quality sepsis care. This study tests interruptive (pop-up) EHR alerts. Epic Systems, the company that produces the EHR, refers to these types of alerts as BestPractice Advisories (BPAs).

ELIGIBILITY:
Patient Inclusion Criteria:

* age > 18 years-old
* meets SIRS criteria
* physically located in the emergency department
* not located in a hospital unit that takes care of pregnant and peri-partum patients
* not SARS-COV-2 PCR positive in past 7 days
* does not have an active order for "comfort measures only"

Patient Exclusion Criteria:

* already having sepsis treatment ordered (if prescribing clinician alert) or collected/completed (if nurse alert)
* already enrolled in the SEPTIC study (including as an emergency department patient or as an inpatient)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25668 (Actual)
Dates: Start 2023-11-14 (Actual); Primary Completion 2024-04-22 (Actual); Study Completion 2024-07-22 (Actual)

PRIMARY OUTCOMES:
Percentage of patients treated with Surviving Sepsis Campaign (SSC) hour-1 bundle | Up to 3 hours
  The primary outcome is whether a patient receives a modified SSC hour-1 bundle within three hours from the time of first SIRS alert. The modified SSC hour-1 bundle includes (1) lactate lab collected, (2) two blood cultures collected, (3) new intravenous antimicrobial administration (from the Centers for Disease Control and Prevention (CDC) Adult Sepsis Event (ASE) list). Patients will be tallied.

SECONDARY OUTCOMES:
Time to blood culture order | 24 hours
  Time from the first SIRS alert until two blood cultures ordered in all patients and the subgroups of patients with CDC ASE, CDC BSE, and Sepsis-3 sepsis definitions. This will be measured in minutes.
Time to blood culture collection | 24 hours
  Time from the first SIRS alert until two blood cultures collected in all patients and the subgroups of patients with CDC ASE, CDC BSE, and Sepsis-3 sepsis definitions. This will be measured in minutes.
Time to lactate order | 24 hours
  Time from the first SIRS alert until lactate lab ordered in all patients and the subgroups of patients with CDC ASE, CDC BSE, and Sepsis-3 sepsis definitions. This will be measured in minutes.
Time to lactate collection | 24 hours
  Time from the first SIRS alert until lactate lab collected in all patients and the subgroups of patients with CDC ASE, CDC BSE, and Sepsis-3 sepsis definitions. This will be measured in minutes.
Time to antibiotic order | 24 hours
  Time from the first SIRS alert until new antibiotic order in all patients and the subgroups of patients with CDC ASE, CDC BSE, and Sepsis-3 sepsis definitions. This will be measured in minutes.
Time to antibiotic treatment | 24 hours
  Time from the first SIRS alert until new antibiotic administration in all patients and the subgroups of patients with CDC ASE, CDC BSE, and Sepsis-3 sepsis definitions. This will be measured in minutes.
Sepsis incidence | Up to 90 days
  Sepsis incidence (CDC ASE, CDC BSE, Sepsis-3) across all alerting groups. Events will be recorded and tallied up to 90 days from first SIRS alert or discharge, whichever occurs first.
Percentage of patients transferred to ICU transfer | Up to 90 days
  Intensive care unit (ICU) transfers for patients not in the ICU at the time of first SIRS alert will be recorded and tallied up to 90 days from first SIRS alert or discharge, whichever occurs first.
Median number of days of hospitalization | Up to 90 days
  This is to determine the average length of stay in the hospital. Days will be recorded and tallied up to 90 days from first SIRS alert or discharge, whichever occurs first.
Percentage of patients discharged as deceased or discharged to hospice | Up to 90 days
  This is to measure the outcomes ended in death or hospice. Outcomes will be recorded and tallied up to 90 days from first SIRS alert or discharge, whichever occurs first.
Percentage of patients discharged home | Up to 90 days
  This is to measure the outcomes ended in returning to home. Outcomes will be recorded and tallied up to 90 days from first SIRS alert or discharge, whichever occurs first.
Percentage of patients discharged to rehab | Up to 90 days
  This is to measure the outcomes ended in rehab. Outcomes will be recorded and tallied up to 90 days from first SIRS alert or discharge, whichever occurs first.
Percentage of patients discharged to skilled nursing facility | Up to 90 days
  This is to measure the outcomes ended in skilled nursing facility. Outcomes will be recorded and tallied up to 90 days from first SIRS alert or discharge, whichever occurs first.
Percentage inpatient mortality at 90 days | Up to 90 days
  This is to measure inpatient mortality. Deaths will be recorded and tallied up to 90 days from first SIRS alert or discharge, whichever occurs first.
Number of positive blood cultures | Up to 90 days
  Positive blood cultures will be determined by blood tests. Positive cultures will be recorded and tallied up to 90 days from first SIRS alert or discharge, whichever occurs first.
Adverse antibiotic events | Up to 90 days
  This is defined as new antibiotic allergy documented in 14 days after first SIRS alert or C. difficile infection or multi-drug resistant organism infection within 7-90 days of first SIRS alert. Events will be recorded and tallied up to 90 days from first SIRS alert or discharge, whichever occurs first.
Time to modified SSC hour-1 bundle completion | 24 hours
  Time interval from first SIRS alert to a modified SSC hour-1 bundle completion, censored at 24 hours after the first alert time, in all patients and the subgroups of patients with CDC ASE, CDC Bacteraemia/Fungemia Shock Event (BSE), and Sepsis-3 sepsis definitions. This will be measured in minutes.

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin L Ranard, MD, MSHP, Study Director — Columbia University; Jason S Adelman, MD, MS, Principal Investigator — Columbia University
Locations (1):
- NewYork-Presbyterian Hospitals, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ranard BL, Qian M, Cummings MJ, Zhang DY, Lee SM, Beitler JR, Applebaum JR, Schenck EJ, Mohamed H, Trepp R, Hsu H, Scofi J, Southern WN, Rossetti SC, Yip NH, Brodie D, Sharma M, Fertel BS, Adelman JS. Pragmatic, multicentre, factorial, randomised controlled trial of sepsis electronic prompting for timely intervention and care (SEPTIC trial): a protocol. BMJ Open. 2025 Aug 11;15(8):e088792. doi: 10.1136/bmjopen-2024-088792. PMID 40789731